CLINICAL TRIAL: NCT01926522
Title: Technological Rehabilitation of Distal Sensorimotor Polyneuropathy in Diabetic
Brief Title: Technological Rehabilitation of Distal Sensorimotor Polyneuropathy in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giovanni Taveggia (Other)
Responsible Party: Sponsor-Investigator, Giovanni Taveggia, MD, Habilita, Ospedale di Sarnico
Organization: Habilita, Ospedale di Sarnico (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Habilita-RAR-02; 201206180007491711110 (Other: Bioethic board)
Record Dates: First submitted 2013-08-14; First posted 2013-08-21 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Complications of Diabetes Mellitus; Diabetic Neuropathies
Keywords: Exercise Therapy
MeSH Terms: conditions — Diabetes Complications; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Technological Rehabilitation (Experimental): Experimental group receives a treatment of: 20 minutes of analyzing treadmill with feedback focused on symmetry and length of stride; 20 minutes of isokinetic dynamometric muscle strengthening of flexor and extensor muscles of tibiotarsal joint; 20 minutes of balance retraining on dynamic balance platform. Each patient receives 20 sessions over a period of 4 weeks (5 sessions per week).
  Interventions: Device: Technological Rehabilitation
- Control Rehabilitation (Active Comparator): Control group receives the same number of treatment sessions of same duration as those in the experimental group: activities targeted to improve the endurance (instead of analyzing treadmill ), manual exercises of lower limb muscle strengthening, stretching exercises (instead of dynamometer), gait retraining on the floor for 20 minutes and static and dynamic balance exercises in upright position (instead of dynamic balance platform).
  Interventions: Other: Control Rehabilitation

INTERVENTIONS:
Device: Technological Rehabilitation — The length of stride of reference used during the exercise is personalized and depends on the height of patients. Each patient carries out the feedback for 20 minutes with the aim of generating the most symmetric and regular gait.
  Patients, with the dynamometer, work on strengthening of flexor and extensor muscles with ankle speeds at 90°/sec and 120°/sec. The strengthening technique was performed twice for 10 minutes each time with a 1 minute rest between sets.
  The session ends with a 20-minute feedback on dynamic balance platform by carrying out exercises in which they need to reach randomly appearing targets. Subjects begin with 12 minutes the first 4 sessions, progress to 16 minutes the next 2 sessions, then 18' (2 sessions), and finally 20', if able, during the last 4 sessions.
  Other Names: Dynamometric isokinetic device: Biodex System 4,; Balance device: Biodex Balance System SD,; Analyzing treadmill: Biodex Gait Trainer 3.
  Arms: Technological Rehabilitation
Other: Control Rehabilitation — When needed, more than on e therapist are employed in the intervention for safety reasons.
  Other Names: Manual rehabilitation with the therapist.
  Arms: Control Rehabilitation

SUMMARY:
The investigators evaluated the effectiveness of the application of analysing treadmill, muscle strengthening and balance training compared to a control intervention in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
Recent studies witnessed how physical exercise may interrupt the devastating decrease of muscle performance in DSP and further experiments are underway to find more exercises for the recovery of motor function impairment. In fact the rehabilitation treatment, that aims at reducing motor disability, preserving gait functions and preventing falling risks, is an interesting therapeutic approach. Literature recommends balance re-training exercises, muscle strengthening, selective stretching and retraining of motor activity.

New technologies produced in the recent decades different devices used in strengthening exercises (electromechanical dynamometers), balance recovery (balance platforms) and gait (analyzing treadmills) have visual feedbacks through which the patients may independently monitor accuracy and intensity of their exercises, being therefore strongly motivated and resulting in a high training intensity. These technologies are often used in rehabilitation of different patients, but are rarely employed for DSP.

The purpose of this case control study was to examine the effectiveness of the application of analysing treadmill, muscle strengthening and balance training compared to a control intervention in patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* The participants need to have a history of diabetes mellitus type 2, >3 years, (i.e., time from the diagnosis or the beginning of first related signs or symptoms),
* A diagnosis of Distal Sensorimotor Polyneuropathy associated,
* Able to walk autonomously, eventually with a aid.

Exclusion Criteria:

* Scoring less than 5 points on the Functional Independence Measure (FIM) (7) locomotion scale,
* Presenting articular ankyloses, contractures, spasms with important locomotion effects,
* Presenting bony instability affecting lower limb functionality (unconsolidated fractures, vertebral instability, severe osteoporosis),
* In presence of attendant clinicopathological conditions contraindicating the rehabilitation treatment (respiratory insufficiency, cardiac/circulatory failure, osteomyelitis, phlebitis and different other conditions),
* In presence of cutaneous lesions at lower limbs,
* Scoring less than 22 points on the Mini Mental State Examination (MMSE),
* Exhibit important behavioural diseases involving aggressivity or psychotic disorders.
* Had received prior interventions for Distal Sensorimotor Polyneuropathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of 6-minute walk test | 1 day after the treatment
  All evaluation procedures are performed by the same examiner who was blinded to the aims of the study and to which group the participants are allocated. The 6-minute walk test (6MWT) is used to assess endurance.
  The 6MWT quantifies functional mobility based on the distance in meters traveled in six minutes. This outcome is a measure of endurance and is particularly significant to evaluate the possibility to perform continuative tasks, that are particularly important for the rehabilitation of diabetic patients and are relevant for an autonomous life. Subjects are instructed to walk at a comfortable speed and subjects neurological are able to use assistive devices.
Change from Baseline of 10-metres walk test | 1 day after the treatment
  All evaluation procedures are performed by the same examiner who was blinded to the aims of the study and to which group the participants are allocated. The 10-metres walking test is used to assess gait speed.
  The speed is quantified with the 10-metres walk test (TWT) over the ground. The gait speed measurement is performed over the middle 6 meters of the TWT and patients are asked to walk at their comfortable speed. Subjects are instructed to walk at a comfortable speed and subjects neurological are able to use assistive devices.

SECONDARY OUTCOMES:
Followup change from Baseline of 6-minute walk test | 30 days after the treatment
  All evaluation procedures are performed by the same examiner who was blinded to the aims of the study and to which group the participants are allocated. The 6-minute walk test (6MWT) is used to assess endurance.
  The 6MWT quantifies functional mobility based on the distance in meters traveled in six minutes. This outcome is a measure of endurance and is particularly significant to evaluate the possibility to perform continuative tasks, that are particularly important for the rehabilitation of diabetic patients and are relevant for an autonomous life. Subjects are instructed to walk at a comfortable speed and subjects neurological are able to use assistive devices.
Followup change from Baseline of 10-metres walk test | 30 days after the treatment
  All evaluation procedures are performed by the same examiner who was blinded to the aims of the study and to which group the participants are allocated. The 10-metres walking test is used to assess gait speed.
  The speed is quantified with the 10-metres walk test (TWT) over the ground. The gait speed measurement is performed over the middle 6 meters of the TWT and patients are asked to walk at their comfortable speed. Subjects are instructed to walk at a comfortable speed and subjects neurological are able to use assistive devices.
Change from Baseline of the Functional Independence Measure (FIM) | 1 day after the treatment
Change from Baseline of the Tinetti scale | 1 day after the treatment
Change from Baseline of the Resting Energy Expenditure (REE) | 1 day after the treatment
Change from Baseline of the Respiratory Rate (RR) | 1 day after the treatment
Change from Baseline of the Heart Rate (HR) | 1 day after the treatment
Change from Baseline of the oxygen saturation (SpO2) | 1 day after the treatment
Change from Baseline of the maximal oxygen consumption (VO2 max) | 1 day after the treatment
Change from Baseline of the expired minute volume (Ve) | 1 day after the treatment
Change from Baseline of the fraction of expired air that is oxygen (FeO2) | 1 day after the treatment
Change from Baseline of the Systolic Blood Pressure (SBP) | 1 day after the treatment
Change from Baseline of the Diastolic Blood Pressure (DBP) | 1 day after the treatment
Change from Baseline of the Glycated Hemoglobin (HbA1c) | 1 day after the treatment
Followup change from Baseline of the Functional Independence Measure (FIM) | 30 days after the treatment
Followup change from Baseline of the Tinetti scale | 30 days after the treatment
Followup change from Baseline of the Resting Energy Expenditure (REE) | 30 days after the treatment
Followup change from Baseline of the Respiratory Rate (RR) | 30 days after the treatment
Followup change from Baseline of the Heart Rate (HR) | 30 days after the treatment
Followup change from Baseline of the oxygen saturation (SpO2) | 30 days after the treatment
Followup change from Baseline of the maximal oxygen consumption (VO2 max) | 30 days after the treatment
Followup change from Baseline of the expired minute volume (Ve) | 30 days after the treatment
Followup change from Baseline of the fraction of expired air that is oxygen (FeO2) | 30 days after the treatment
Followup change from Baseline of the Systolic Blood Pressure (SBP) | 30 days after the treatment
Followup change from Baseline of the Diastolic Blood Pressure (DBP) | 30 days after the treatment
Followup change from Baseline of the Glycated Hemoglobin (HbA1c) | 30 days after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Taveggia, MD, Principal Investigator — Habilita, Ospedale di Sarnico
Locations (1):
- Habilita, Ospedale di Sarnico, Sarnico, Bergamo, Italy

REFERENCES:
- [Background] Andersen H. Motor dysfunction in diabetes. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:89-92. doi: 10.1002/dmrr.2257. PMID 22271730
- [Background] Starling JR, Harms BA. Diagnosis and treatment of genitofemoral and ilioinguinal neuralgia. World J Surg. 1989 Sep-Oct;13(5):586-91. doi: 10.1007/BF01658875. PMID 2815802
- [Background] Ites KI, Anderson EJ, Cahill ML, Kearney JA, Post EC, Gilchrist LS. Balance interventions for diabetic peripheral neuropathy: a systematic review. J Geriatr Phys Ther. 2011 Jul-Sep;34(3):109-16. doi: 10.1519/JPT.0b013e318212659a. PMID 21937901
- [Background] Fedele D, Comi G, Coscelli C, Cucinotta D, Feldman EL, Ghirlanda G, Greene DA, Negrin P, Santeusanio F. A multicenter study on the prevalence of diabetic neuropathy in Italy. Italian Diabetic Neuropathy Committee. Diabetes Care. 1997 May;20(5):836-43. doi: 10.2337/diacare.20.5.836. PMID 9135952
- [Background] Aring AM, Jones DE, Falko JM. Evaluation and prevention of diabetic neuropathy. Am Fam Physician. 2005 Jun 1;71(11):2123-8. PMID 15952441
- [Background] Divisova S, Vlckova E, Hnojcikova M, Skorna M, Nemec M, Dubovy P, Dusek L, Jarkovsky J, Belobradkova J, Bednarik J. Prediabetes/early diabetes-associated neuropathy predominantly involves sensory small fibres. J Peripher Nerv Syst. 2012 Sep;17(3):341-50. doi: 10.1111/j.1529-8027.2012.00420.x. PMID 22971096
- [Background] Spencer RJ, Wendell CR, Giggey PP, Katzel LI, Lefkowitz DM, Siegel EL, Waldstein SR. Psychometric limitations of the mini-mental state examination among nondemented older adults: an evaluation of neurocognitive and magnetic resonance imaging correlates. Exp Aging Res. 2013;39(4):382-97. doi: 10.1080/0361073X.2013.808109. PMID 23875837
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Bennell K, Dobson F, Hinman R. Measures of physical performance assessments: Self-Paced Walk Test (SPWT), Stair Climb Test (SCT), Six-Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S350-70. doi: 10.1002/acr.20538. No abstract available. PMID 22588756
- [Background] Nascimento LR, Caetano LC, Freitas DC, Morais TM, Polese JC, Teixeira-Salmela LF. Different instructions during the ten-meter walking test determined significant increases in maximum gait speed in individuals with chronic hemiparesis. Rev Bras Fisioter. 2012 Apr;16(2):122-7. doi: 10.1590/s1413-35552012005000008. Epub 2012 Mar 1. English, Portuguese. PMID 22378478
- [Background] Gomes AA, Onodera AN, Otuzi ME, Pripas D, Mezzarane RA, Sacco IC. Electromyography and kinematic changes of gait cycle at different cadences in diabetic neuropathic individuals. Muscle Nerve. 2011 Aug;44(2):258-68. doi: 10.1002/mus.22051. PMID 21755508
- [Background] van Sloten TT, Savelberg HH, Duimel-Peeters IG, Meijer K, Henry RM, Stehouwer CD, Schaper NC. Peripheral neuropathy, decreased muscle strength and obesity are strongly associated with walking in persons with type 2 diabetes without manifest mobility limitations. Diabetes Res Clin Pract. 2011 Jan;91(1):32-9. doi: 10.1016/j.diabres.2010.09.030. Epub 2010 Oct 20. PMID 20965601
- [Background] Thomas T, Schreiber G. Acute-phase response of plasma protein synthesis during experimental inflammation in neonatal rats. Inflammation. 1985 Mar;9(1):1-7. doi: 10.1007/BF00915406. PMID 2579907
- [Background] Corriveau H, Prince F, Hebert R, Raiche M, Tessier D, Maheux P, Ardilouze JL. Evaluation of postural stability in elderly with diabetic neuropathy. Diabetes Care. 2000 Aug;23(8):1187-91. doi: 10.2337/diacare.23.8.1187. PMID 10937520